CLINICAL TRIAL: NCT06256380
Title: Comparing Enhanced Cognitive-behavior Therapy and Family-based Treatment for Adolescents With an Eating Disorder: a Non-inferiority Randomized Controlled Trial
Brief Title: Comparing Enhanced Cognitive-behavior Therapy and Family-based Treatment for Adolescents With an Eating Disorder
Acronym: CogFam
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other); University of Oslo (Other); Villa Garda Hospital (Other); University of California, San Francisco (Other); St. Olavs Hospital (Other); University Hospital of North Norway (Other); Haukeland University Hospital (Other); Vestre Viken Hospital Trust (Other)
Responsible Party: Principal Investigator, Øyvind Rø MD, Research director, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CogFamNorway
Record Dates: First submitted 2023-12-21; First posted 2024-02-13 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Feeding and Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced cognitive-behavior therapy for adolescents with an eating disorder (CBT-E) (Experimental): CBT-E posits the eating problem as belonging to the individual, and is designed to encourage the adolescent, rather than their parent, to take control of the problem. Parents are not excluded from participating in treatment, but their involvement is limited to helping to create a family environment that allows for recovery. Patients are actively involved in all phases of treatment, including the decision to address weight regain and/or binge eating and purging, with the goal of promoting self-management. A primary goal of CBT-E is to address the patient's eating disorder psychopathology, i.e. patients' concerns about shape, weight, dietary restraint and restriction, and other extreme weight control behaviors. Following manualized CBT-E guidelines, for patients in the lower weight cohort, treatment involves 40 sessions over 9-12 months. For those in the higher weight cohort, treatment involves 20 sessions over the course of 6 months.
  Interventions: Behavioral: Enhanced Cognitive-behavior therapy for adolescents with an eating disorder
- Family-based treatment for adolescents with an eating disorder (FBT) (Active Comparator): FBT for adolescent eating disorders usually includes all members of the adolescent's immediate family. Treatment progresses through three phases, with the first (∼10 sessions) focusing mainly on guiding the parents to support their adolescent toward weight restoration (when appropriate), and disrupting eating disorder behaviors (e.g. binge eating and purging). The second phase (∼5-7 sessions) focuses on assisting the parents to restore food choices to the adolescent, with an emphasis on the developmental stage of the adolescent. Phase 3 is brief (2-3 sessions), focusing on adolescent developmental matters and helping the parents and their offspring navigate these tasks largely in the absence of acute eating disorder symptoms. Twenty treatment sessions are provided over a span of approximately 6 months.
  Interventions: Behavioral: Family-based therapy for adolescents with an eating disorder

INTERVENTIONS:
Behavioral: Enhanced Cognitive-behavior therapy for adolescents with an eating disorder — Psychotherapy
  Arms: Enhanced cognitive-behavior therapy for adolescents with an eating disorder (CBT-E)
Behavioral: Family-based therapy for adolescents with an eating disorder — Psychotherapy
  Arms: Family-based treatment for adolescents with an eating disorder (FBT)

SUMMARY:
The goal of this randomized controlled clinical trial is to compare the efficacy of outpatient family-based treatment versus enhanced cognitive behavior therapy for children and adolescents with eating disorders.

Because of insufficient recruitment, the study design was modified on December 1st, 2025, to a partially randomized preference design.

The main aim is to determine if enhanced cognitive behavior therapy has a similar efficacy as family-based treatment among children and adolescents with eating disorders receiving treatment in an outpatient setting. The main outcome is improvement in eating disorders psychopathology at the end of treatment.

DETAILED DESCRIPTION:
Eating disorders (EDs) are severe mental illnesses, associated with high morbidity, increased mortality, and reduced quality of life. Despite treatment advancements, remission rates are modest. Even in specialized treatment settings offering evidence-based treatments such as family-based treatment (FBT), remission rates are about 50%. There is emerging evidence for the effectiveness of enhanced cognitive behavior therapy (CBT-E) for adolescents with EDs. However, no randomized controlled trial (RCT) has yet compared these two treatments.

The current study will compare FBT, which has proven efficacious and is currently recommended for adolescents with EDs, and the newer treatment approach of CBT-E in a large, national RCT. Young patients with all EDs (12-18 years of age) undergoing outpatient treatment from eight different clinics in Norway will be invited to participate in the study.

Because of insufficient recruitment, the study design was modified on December 1st, 2025, to a partially randomized preference design.

Primary aim:

This study is a randomized controlled trial comparing the efficacy of outpatient family-based treatment versus enhanced cognitive behavior therapy for children and adolescents with eating disorders. The main outcome is improvement in eating disorders psychopathology at the end of treatment.

Secondary aims:

To compare weight gain for underweight patients, changes in comorbid psychopathology including depression, self-esteem, family functioning, and quality of life at 6-and 12-months follow-up.

Potential moderators of outcome will be explored. Treatment satisfaction and experiences of the two different treatments will be investigated from the perspective of patients, parents, and clinicians. Data from the Norwegian Control and Payment of Health Reimbursements Database (KUHR), the Norwegian Patient Registry (NPR), and Social Security Database will be obtained to compare the direct and indirect costs of health care utilization for the two treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnosed eating disorder
2. Medically stable for outpatient treatment.
3. Living with at least one of their parents
4. At least one of their parents could be actively involved in the treatment
5. Sufficient knowledge in reading, understanding and speaking Norwegian

Exclusion Criteria:

1. Avoidant restrictive food intake disorders
2. A co-morbid medical condition or disorder known to influence eating or weight, or influence the possibilities to take part in treatment
3. Psychotic disorders
4. Acute suicidality
5. Substance abuse and/or substance dependence
6. Serious traumatic events in the family making treatment following FBT or CBT-E manual not recommended
7. Unstable psychotropic medication last 6 weeks

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in eating disorder psychopathology | Baseline, immediately after the intervention.
  Change in global scores on a well-validated semi-structured interview of eating disorder attitudes and behavior, the Eating Disorder Examination - Interview. Possible scores range from 0-6 where higher scores indicate worse symptoms.

SECONDARY OUTCOMES:
Change in eating disorder psychopathology | Baseline, immediately after the intervention, 6 months after the end of treatment, 12 months after the end of treatment.
  Change in global and subscale scores on a well-validated self-report questionnaire of eating disorder attitudes and behavior, the Eating Disorder Examination-Questionnaire. Possible scores range from 0-6 where higher scores indicate worse symptoms.
Change in weight (kg) for underweight participants (defined as those participants who are below 18,5 Body Mass Index (BMI) (kg/m2) at baseline or corresponding BMI to age and gender). | Baseline, immediately after the intervention, 6 months after the end of treatment, 12 months after the end of treatment
  Weight gain in kilogram. Higher weight gain means better outcome.
Change in depression | Baseline, immediately after the intervention, 6 months after the end of treatment, 12 months after the end of treatment
  Change in global score on a well-validated self-report questionnaire of depression, the Beck Depression Inventory II. Possible scores range from 0 to 63 where higher scores mean worse symptoms.
Change in anxiety | Baseline, immediately after the intervention, 6 months after the end of treatment, 12 months after the end of treatment
  Change in global score on a well-validated self-report questionnaire of anxiety, the Beck Anxiety Inventory. Possible scores range from 0 to 63 where higher scores mean worse symptoms.
Change in quality of life | Baseline, immediately after the intervention, 6 months after the end of treatment, 12 months after the end of treatment
  Change in global score on a well-validated self-report measure of quality of life, Health-Related Quality of Life Index (KIDDIESCREEN 10). Possible scores range from 10 to 50 where higher scores mean better quality of life.
Change in impairment due to eating difficulties | Baseline, immediately after the intervention, 6 months after the end of treatment, 12 months after the end of treatment
  Change in global score on well validated self report measure of eating disorders-specific quality of life, the Clinical Impairment assessment. Possible scores range from 0 (no impairment) to 48 (highest level of impairment).
Change in self-esteem | Baseline, immediately after the intervention, 6 months after the end of treatment, 12 months after the end of treatment
  Change in global score on a well validated self-report measure of self-esteem, the Rosenberg Self-Esteem Scale questionnaire. Scores range from 10 to 40, where higher scores mean better self-esteem.

OTHER OUTCOMES:
Changes in family function | Baseline, immediately after the intervention, 6 months after the end of treatment, 12 months after the end of treatment
  Change in parent ratings of family functioning measured by the subscale score on a well validated self-report questionnaire- the McMaster Family Assessment Device, General Functioning subscale. Scores on this subscale range from 12 to 48, where higher scores means worse level of family function.
Changes caregiving experience and psychological symptoms | Baseline, immediately after the intervention, 6 months after the end of treatment, 12 months after the end of treatment
  Change in parent ratings on the impact of eating disorder symptoms on caregiving experiences measured by a well validated, self-report measure -the Eating Disorders Symptom Impact Scale. Scores range from 0 to 96, where higher scores mean worse impact of eating disorder symptoms.
Changes caregiving mental health | Baseline, immediately after the intervention, 6 months after the end of treatment, 12 months after the end of treatment
  Change in parent ratings on the mental health symptoms by a well validated, self-report measure -the Hopkins symptoms checklist 25 items. Scores range from 1 to 4 where higher scores mean worse mental health symptoms.
Direct and indirect costs of health care use for patients and parents/caregivers | Baseline, immediately after the intervention, 6 months after the end of treatment, 12 months after the end of treatment
  Register data from the Norwegian Control and Payment of Health Reimbursements Database (KUHR), the Norwegian Patient Registry (NPR), and Social Security Database.

CONTACTS AND LOCATIONS:
Overall Officials: Øyvind Rø, MD, Principal Investigator — Oslo University Hospital; Ingrid Funderud, PhD, Principal Investigator — Oslo University Hospital
Locations (5):
- Norway (5):
  - Haukeland University Hospital, Bergen
  - Vestre Viken Health Trust, Drammen
  - Oslo University Hospital, Oslo
  - University Hospital of North Norway, Tromsø
  - St. Olav Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No